CLINICAL TRIAL: NCT06619704
Title: A rEtrospectIve Real-world Analysis of earLy responsE ratEs With Ribociclib and Endocrine Therapy and Descriptive aNalysis of HR+, HER2- Metastatic Breast Cancer Patients Treated With Chemotherapy (EILEEN)
Brief Title: Observational Retrospective Study to Assess the Use of Ribociclib in Patients With HR+, HER2- Metastatic Breast Cancer Treated With Chemotherapy
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011ATR01
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Group I: Postmenopausal female patients who initiated ribociclib combinations per local label.
- Group II: Postmenopausal female patients who were eligible for cyclin-dependent kinase inhibitors (CDKis) according to local label but started chemotherapy.

SUMMARY:
EILEEN was a non-interventional/observational, retrospective, multi-center, real life cohort study conducted in 14 private and academic oncology clinics in Turkey. Group I cohort of the study was based on secondary use of data of postmenopausal hormone receptor-positive (HR+), human epidermal growth factor receptor 2-negative (HER2-) metastatic breast cancer (MBC) patients treated with ribociclib in combination with letrozole (LET) or fulvestrant (FUL) after June 2020. Group II cohort of the study was a parallel, comprehensive chart review for detecting all postmenopausal HR+, HER2- MBC patients who were eligible for cyclin-dependent kinase inhibitors (CDKis) but received chemotherapy. The study used secondary data which was retrieved from electronic or paper medical records or clinical databases available at the sites. Regular follow up with close monitorization was used for the effective management of patients with breast cancer. Data sources included information about diagnosis, treatment and monitorization of patients at an individual level. The study used medical patient records at hospitals e.g. hospital discharge files, primary clinical records and electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

Group I: Postmenopausal female patients who had histologically or cytologically confirmed HR-positive (10% or more ER+), HER2-negative, metastatic breast cancer and initiated ribociclib combinations per local label.

* Treated with ribociclib plus letrozole relapsed after 12 months completing adjuvant treatment or without any prior endocrine treatment for metastatic disease, 1 line or less chemotherapy was allowed.
* Treated with ribociclib plus fulvestrant, clinical and/or radiological disease progression after at least 6 months and at least 1 aromatase inhibitor treatment for metastatic disease or relapsed after 12 months adjuvant aromatase inhibitor treatment and/or relapsed within 12 months completing adjuvant aromatase inhibitor, 2 lines or less prior treatments and 1 line or less prior chemotherapy at metastatic setting were allowed.
* Had first treatment response rate assessment within 6 months after ribociclib initiation.
* Initiated ribociclib in combination with letrozole/fulvestrant after MBC diagnosis after local approval of ribociclib in June 2020.

Group II: Postmenopausal female patients who had histologically or cytologically confirmed HR-positive (10% or more ER+), HER2-negative, metastatic breast cancer eligible for cyclin-dependent kinase (CDK) inhibitors according to local label but started chemotherapy.

Exclusion Criteria:

* Pre- or perimenopausal women.
* Enrollment in an interventional clinical trial for MBC during the study observation period.
* Evidence of prior treatment with any CDK4/6 inhibitor in the adjuvant setting.
* Evidence of another primary cancer within 3 years prior to the initial line containing ribociclib.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal female patients who had histologically or cytologically confirmed HR-positive (10% or more estrogen receptor-positive [ER+]), HER2-negative, metastatic breast cancer
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) at First Assessment After Initiation of Treatment Combinations | Up to 6 months
  Treatment combinations included ribociclib plus letrozole and ribociclib plus fulvestrant.
  ORR was defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR) according to RECIST v1.1.

SECONDARY OUTCOMES:
Number of Patients Categorized by Former Treatment | Baseline
Number of Patients who Used Chemotherapy per Treatment Combination | Up to 3 years
  Treatment combinations included ribociclib plus letrozole and ribociclib plus fulvestrant.
Progression Free Survival (PFS) | Up to 3 years
  PFS was defined as the time from date of start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient did not have an event, PFS was censored at the date of last adequate tumor assessment.
Overall Survival (OS) | Up to 3 years
  OS was defined as the time from date of start of treatment to date of death due to any cause. If a patient was not known to have died, survival was censored at the date of last known date patient was alive.
Time to Progression | Up to 3 years
Time to Chemotherapy Post-ribociclib Plus Letrozole or Fulvestrant Treatments | Up to 3 years
Duration of Treatment | Up to 3 years
Proportion of Patients With Complete Response (CR)/Partial Response (PR)/Stable Disease (SD)/Progressive Disease (PD) | Up to 6 months
  CR was defined as the disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have had a reduction in short axis to less than 10 mm.
  PR was defined as at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
  SD was defined as neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD.
  PD was defined as at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must have also demonstrated an absolute increase of at least 5 mm.
Clinical Benefit Rate (CBR) | Up to 6 months
  Clinical benefit rate: ORR and as defined by RECIST 1.1. CBR was defined as percentage of patients with complete response (CR), partial response (PR) per RECIST or stable disease (SD) lasting 24 weeks or longer.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States